CLINICAL TRIAL: NCT03005925
Title: An Open Prospective Randomized Controlled Study Comparing the Use of Remote Monitoring by Smartphone in the Care Management of Patients With Rheumatoid Arthritis Versus a Standard Outpatient Follow-up by Physical Consultation
Brief Title: Use of Remote Monitoring by Smartphone in the Care Management of Patients With Rheumatoid Arthritis
Acronym: SATIE-PR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: European Union (Other); Occitanie Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL_0174
Record Dates: First submitted 2016-12-19; First posted 2016-12-30 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- connected group (Experimental): remote monitoring by smartphone in the care management of patients with rheumatoid arthritis
  Interventions: Device: Smartphone
- control group (Active Comparator): standard outpatient follow-up by physical consultation
  Interventions: Other: physical follow up

INTERVENTIONS:
Device: Smartphone — Smartphone application coupled with a hand dynamometer
  Other Names: tele medicine follow up
  Arms: connected group
Other: physical follow up — regular visits with the specialist
  Arms: control group

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatism in adults, affecting nearly 0.4% of the general population. It is a real public health issue. International guidelines recommend strict control (remission or low disease activity) of the disease, to avoid joint destruction in order to reduce the functional impact of the disease in the long term and to improve the quality of life of the patients.

This care is based on a close follow-up requiring regular visits with the specialist which represents an additional cost (transport, visits). In this context, tele-medicine is often proposed as a complementary approach in the management of these chronic patients.

Thus, the investigators propose to study the interest of a connected device by comparing a group of patients using this Smartphone application, coupled with a hand dynamometer during the 6 months following initiation of a new DMARD.

ELIGIBILITY:
Inclusion Criteria:

* • Patients between 18 and 75 years old with rheumatoid arthritis according to 2010 ACR (American College of Rheumatology) / EULAR Classification Criteria

  * Patients that need a treatment initiation for rheumatoid arthritis
  * Patients with DAS 28 > 3.2 (Disease Activity Score )
  * Patients who agreed to participate in this study and provide the informed consent

Exclusion Criteria:

* • Insufficient level of understanding to perform the measurement and self-report questionnaires

  * Patients without an internet connection
  * Difficulties in using a dynamometer due to a dominant-hand surgery done during the previous 12 months, carpal tunnel symptoms, or ulnar nerve compression, or cervicobrachial neuralgia, known presence of motor dysfunction of the upper extremity, or neurological disease
  * Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Consultation | follow up of patients over 6 months
  To evaluate whether the use of a computerized monitoring interface on Smartphone ( "SATIE-PR" application) reduces the number of consultations during follow-up of patients with RA over 6 months
Number of consultations | follow up of patients over 6 months
  % of patients who benefit from at least 4 consultations over a 6-month period.

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pers YM, Valsecchi V, Mura T, Aouinti S, Filippi N, Marouen S, Letaief H, Le Blay P, Autuori M, Fournet D, Mercier G, Ferreira R, Jorgensen C. A randomized prospective open-label controlled trial comparing the performance of a connected monitoring interface versus physical routine monitoring in patients with rheumatoid arthritis. Rheumatology (Oxford). 2021 Apr 6;60(4):1659-1668. doi: 10.1093/rheumatology/keaa462. PMID 33020846
- [Derived] Bernard L, Valsecchi V, Mura T, Aouinti S, Padern G, Ferreira R, Pastor J, Jorgensen C, Mercier G, Pers YM. Management of patients with rheumatoid arthritis by telemedicine: connected monitoring. A randomized controlled trial. Joint Bone Spine. 2022 Oct;89(5):105368. doi: 10.1016/j.jbspin.2022.105368. Epub 2022 Mar 4. PMID 35248737